CLINICAL TRIAL: NCT01443897
Title: Effect of Consumption of Post-harvest UV-B Treated Mushrooms on Vitamin D Status of Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 201017924-1
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Placebo Comparator): Untreated mushrooms plus placebo capsule.
  Interventions: Dietary Supplement: placebo capsule; Other: mushrooms
- Group 2 (Experimental): UVB-treated mushrooms (400 IU vitamin D2 per serving) plus placebo capsule.
  Interventions: Dietary Supplement: placebo capsule; Other: UVB-treated mushrooms, 400 IU vitamin D2
- Group 3 (Experimental): UVB-treated mushrooms (1,000 IU vitamin D2 per serving) plus placebo capsule.
  Interventions: Dietary Supplement: placebo capsule; Other: UVB-treated mushrooms, 1,000 IU vitamin D2
- Group 4 (Experimental): Untreated mushrooms plus 1,000 IU Vitamin D2 in capsule
  Interventions: Dietary Supplement: 1,000 IU vitamin D2; Other: mushrooms

INTERVENTIONS:
Dietary Supplement: 1,000 IU vitamin D2 — capsule containing 1,000 IU vitamin D2
  Arms: Group 4
Dietary Supplement: placebo capsule — 0 IU vitamin D2
  Arms: Group 1; Group 2; Group 3
Other: mushrooms — untreated button mushrooms, obtained from Monterey Mushrooms, Monterey, CA
  Arms: Group 1; Group 4
Other: UVB-treated mushrooms, 400 IU vitamin D2 — UVB-treated button mushrooms, 400 IU vitamin D2 per 1/2 cup serving, obtained from Monterey Mushrooms, Monterey, CA
  Arms: Group 2
Other: UVB-treated mushrooms, 1,000 IU vitamin D2 — UVB-treated button mushrooms, 1,000 IU vitamin D2 per 1/c serving, obtained from Monterey Mushrooms, Monterey, CA
  Arms: Group 3

SUMMARY:
This study will investigate whether mushrooms treated with ultraviolet (UV) light to increase their vitamin D2 content are actually a good source of vitamin D when consumed daily with a meal (lunch). The mushrooms will be provided cooked along with a meal which will be a standard, pre-packaged frozen meal. We also hope to learn if the resulting improvement in vitamin D status affects the immune system by decreasing it's level of activation, which may be abnormally elevated in vitamin D deficiency.

DETAILED DESCRIPTION:
Volunteers will be asked to consume a standard meal (lunch) containing one serving of mushrooms daily for six weeks (7 days per week). With the meal, they will also need to take one capsule. The capsule will be either a placebo or will contain vitamin D. The purpose of the vitamin D in the capsule is to determine if the vitamin D from the mushrooms is absorbed as well as vitamin D from a capsule. The total dose of vitamin D that volunteers will receive each day from mushrooms and capsule together will always be the same and will be one of three doses: (1) little or no vitamin D (placebo); (2) 400 IU, which is near the current recommended intake and (3) 1,000 IU, which is up to five-fold higher than the current recommended intake, depending on your age. Both levels of vitamin D are safe. In addition to consuming the meals and taking the capsules, up to 20 mL (4 teaspoons) of blood will be drawn at three times during the study just before the mushroom-containing lunch is provided: (1) at the beginning of the study before the first meal; (3) after three weeks; (3) at the end of the study. The purpose of the blood draw is to measure vitamin D in your blood and to measure the level of activation of your immune system by measuring markers of immune activation.

ELIGIBILITY:
Inclusion Criteria:

* willing to consume a lunch meal 7 days per week for 6 weeks containing mushrooms
* willing to stop eating other sources of mushrooms
* willing to discontinue taking vitamin D and other dietary supplements
* estimated low vitamin D status based on dietary questionnaire, skin reflectance, and sun behavior

Exclusion Criteria:

* women who are pregnant or breastfeeding
* volunteers with anemia
* volunteers with evidence of underlying disease affecting vitamin D metabolism
* volunteers taking medications altering vitamin D metabolism

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in serum Vitamin D2 | 0, 3 and 6 weeks
  Serum vitamin D 2 will be measured in serum.

SECONDARY OUTCOMES:
Change in serum markers of inflammation | 0, 3, and 6 weeks
  Measure serum cytokines, chemokines, and neopterin.

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Stephensen, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States